CLINICAL TRIAL: NCT04050774
Title: Balance Control Mechanisms During Perturbed Standing Across the Lifespan
Brief Title: Standing Balance Control Across the Lifespan
Acronym: BaCoMech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Pieter Meyns, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Projectlifespanbalance2018-001
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Children, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Age group 1 (Experimental): 6-9 years old
  Interventions: Device: Balance boards
- Age group 2 (Experimental): 15-17 years old
  Interventions: Device: Balance boards
- Age group 3 (Experimental): 18 - 24 years old
  Interventions: Device: Balance boards
- Age group 4 (Experimental): 65-80 years old
  Interventions: Device: Balance boards

INTERVENTIONS:
Device: Balance boards — The unstable surface will be created with a balance board consisting of a wooden board mounted on a section of a cylinder, creating an unstable support in the sagittal plane or in the frontal plane. The participants will stand on three balance boards, varying the height of the surface of the board above the point of contact (15, 17 and 19 cm respectively). The radius of the cylinder will kept constant at 24 cm. The standing surface will be 48cm x 48 cm

SUMMARY:
Falls are the leading cause of nonfatal injuries in children and elderly. To understand the causes of falling in these populations, fundamental knowledge of how ageing affects balance control is of utmost importance.

In general, two biomechanical mechanisms allow people to control balance; 1.moving the center of pressure within the base of support using ankle muscle activation; 2.counter-rotating segments around the center of mass. To understand how balance is controlled differently across the lifespan, 4 age groups (each N=20) will be compared to each other; i.e. prepubertal children (6-9y), postpubertal children (15-17y), young adults (18-24y), healthy non-falling older adults (65-80y). .

A force plate platform combined with 3D movement registration will be used to determine the biomechanical balance control strategy across the lifespan during unperturbed and perturbed standing. The innovative but focused scope of this study could provide a breakthrough in our biomechanical understanding of balance control and, in particular, the changes in limitations of balance control in childhood and an ageing (fall-prone) population. The gained fundamental knowledge could lead to unprecedented insights in the causes of falling across the lifespan and in possible targets for intervention.

ELIGIBILITY:
Inclusion Criteria:

* prepubertal children (6-9y)
* postpubertal children (15-18y)
* young adults (18-24y)
* healthy non-falling older adults (65-80y) will be included if they 1) did not experience two or more falls during normal daily activities in the preceding year and 2) have no cognitive impairment (tested with Mini-Mental state examination).

Exclusion Criteria:

1. inability to speak and understand Dutch;
2. inability to maintain independent unsupported stance for 60 seconds;
3. current diagnosis of neurological or sensory disorders;
4. recurrent dizziness;
5. obesity ;
6. a history of orthopaedic disorders;
7. surgical operation of the lower extremity during last two years;
8. use of drugs affecting the CNS or known to affect balance control.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Balance Control; centre of mass acceleration based on 3D movement registration and ground reaction forces | day 1
  Centre of mass acceleration (in kg.m2/s2) (calculations based on; van Dieen JH, van Leeuwen M, Faber GS. Learning to balance on one leg: motor strategy and sensory weighting. J Neurophysiol. 2015;114(5):2967-82.)
Contribution of the ankle strategy to centre of mass acceleration based on 3D movement registration and ground reaction forces | day 1
  The contribution of the ankle strategy (difference between the centre of pressure and the centre of mass (in kg.m2/s2)) to centre of mass acceleration in the sagittal and frontal plane will be calculated based on total body kinematics (SIMI motion - 3D movement registration) and kinetics (AMTI force plate) (calculations based on; van Dieen JH, van Leeuwen M, Faber GS. Learning to balance on one leg: motor strategy and sensory weighting. J Neurophysiol. 2015;114(5):2967-82.)
Contribution of the counter-rotation mechanism to centre of mass acceleration based on 3D movement registration and ground reaction forces | day 1
  The contribution of the counter-rotation mechanism (change in angular momentum (in kg.m2/s2)) to centre of mass acceleration in the sagittal and frontal plane will be calculated based on total body kinematics (SIMI motion - 3D movement registration) and kinetics (AMTI force plate) (calculations based on; van Dieen JH, van Leeuwen M, Faber GS. Learning to balance on one leg: motor strategy and sensory weighting. J Neurophysiol. 2015;114(5):2967-82.))

CONTACTS AND LOCATIONS:
Locations (1):
- Hasselt University, Hasselt, Belgium